CLINICAL TRIAL: NCT01227395
Title: Drug Use Investigation On Zithromac Tablets 600mg In HIV Patients (Post Marketing Commitment Plan)
Brief Title: Drug Use Investigation On Zithromac (Azithromycin) In HIV Patients
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Altmarc Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: A0661097
Record Dates: First submitted 2010-10-07; First posted 2010-10-25 (Estimated); Results first posted 2013-04-16 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: HIV Infection
Keywords: HIV; Post Marketing Surveillance
MeSH Terms: conditions — HIV Infections | interventions — Azithromycin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Azithromycin: Patients taking Azithromycin.
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Inhibition of onset: Perorally administer 1200mg of azithromycin (potency) once a week to adults.
  Treatment: Perorally administer 600mg of azithromycin (potency) once a day to adults.
  Other Names: Zithromac, Zithromax, Azithromycin

SUMMARY:
The investigation will be conducted for the purpose of determining the condition of occurrence of Adverse Events under the actual post-marketing use of Zithromac 600mg Tablet, verifying the therapeutic effects, detecting unknown Adverse Drug Reactions and drug interactions and determining the factors affecting safety and efficacy.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first Zithromac Tablets 600mg should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

Patients need to be administered Zithromac Tablets 600mg in order to be enrolled in the surveillance.

Exclusion Criteria:

Patients not administered Zithromac Tablets 600mg.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects whom an investigator involving A0661097 prescribes the Azithromycin Tablets 600mg (Zithromac Tablets 600mg).
Sampling Method: Probability Sample
Enrollment: 476 (Actual)
Dates: Start 2002-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase 4, observational, open-label study conducted in participants who were prescribed azithromycin by their treating physician per usual clinical practice. Study drug was not provided by the Sponsor.
Groups:
- Azithromycin for Prophylaxis: Participants taking Azithromycin for Prophylaxis according to Japanese Package Insert.
- Azithromycin for Treatment: Participants taking Azithromycin for Treatment according to Japanese Package Insert.
Period: Overall Study
Arm/Group | Azithromycin for Prophylaxis | Azithromycin for Treatment
Started | 391 | 85
Completed | 391 | 84
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin for Prophylaxis | Azithromycin for Treatment | Total
Number analyzed (Participants) | 391 | 84 | 475
Age, Customized [Number; unit: participants]
  <65 years | 381 | 83 | 464
  >=65 years | 10 | 1 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 9 | 40
  Male | 360 | 75 | 435

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Frequency of Treatment Related Adverse Events.
Description: Adverse events mean all unfavorable events that occur in participants after administration of Azithromycin, irrespective of causal relationship to Azithromycin (including clinically problematic abnormal changes in laboratory test values). Treatment related Adverse Events were evaluated in company with the causal relationship to Azithromycin.
Time Frame: 9 years(MAX)
Population: No statistical analysis provided for the frequency of treatment related adverse events.
Measure: Number; unit: participants
Arm/Group | Azithromycin for Prophylaxis | Azithromycin for Treatment
Number analyzed (Participants) | 391 | 84
participants | 73 | 10

2. Primary Outcome: Number of Unlisted Treatment Related Adverse Events in Japanese Package Insert.
Description: Adverse events mean all unfavorable events that occur in participants after administration of Azithromycin, irrespective of causal relationship to Azithromycin (including clinically problematic abnormal changes in laboratory test values). Number of Treatment Related Adverse Events were evaluated in company with the causal relationship to Azithromycin. Unlisted treatment related adverse events were confirmed with listed adverse drug reaction in Japanese package insert.
Time Frame: 9 years(MAX)
Population: No statistical analysis provided for the number of the unlisted treatment related adverse events in Japanese Package Insert.
Measure: Number; unit: Events
Arm/Group | Azithromycin for Prophylaxis | Azithromycin for Treatment
Number analyzed (Participants) | 391 | 84
Events | 37 | 9

3. Primary Outcome: Risk Factors for the Frequency of Treatment Related Adverse Events -Age (Prophylaxis).
Description: Number of participants with Treatment Related Adverse Events(TRAEs) of Azithromycin to determine whether <65 years or >=65 years is significant risk factor.
Time Frame: 9 years(MAX)
Population: The safety analysis population consists of the cases that satisfy the cases conditions and in whom administration of this drug was confirmed.
Measure: Number; unit: participants
Groups:
- <65 Years: Participants with <65 years who taking Azithromycin for Prophylaxis according to Japanese Package Insert.
- >=65 Years: Participants with >=65 years who taking Azithromycin for Prophylaxis according to Japanese Package Insert.
Arm/Group | <65 Years | >=65 Years
Number analyzed (Participants) | 381 | 10
participants | 72 | 1
Statistical Analysis 1: Comparison: <65 Years vs >=65 Years; The risk factor tested was "Age". The null hypothesis is there is no difference between "<65 years and >=65 years " in the frequency of Treatment Related Adverse Events(TRAEs); Test type: Superiority or Other; p = 0.696, Fisher Exact

4. Primary Outcome: Risk Factors for the Frequency of Treatment Related Adverse Events -Gender (Prophylaxis).
Description: Number of participants with Treatment Related Adverse Events(TRAEs) of Azithromycin Tablets to determine whether male or female is significant risk factor.
Time Frame: 9 years(MAX)
Population: as for outcome 3
Measure: Number; unit: participants
Groups:
- Male: Male Participants taking Azithromycin for Prophylaxis according to Japanese Package Insert.
- Female: Female Participants taking Azithromycin for Prophylaxis according to Japanese Package Insert.
Arm/Group | Male | Female
Number analyzed (Participants) | 360 | 31
participants | 65 | 8
Statistical Analysis 1: Comparison: Male vs Female; The risk factor tested was "Gender". The null hypothesis is there is no difference between "Male and Female " in the frequency of Treatment Related Adverse Events(TRAEs); Test type: Superiority or Other; p = 0.334, Fisher Exact

5. Primary Outcome: Risk Factors for the Frequency of Treatment Related Adverse Events -Concomitant Drugs (Prophylaxis).
Description: Number of participants with Treatment Related Adverse Events(TRAEs) of Azithromycin Tablets to determine whether with or without concomitant drugs is significant risk factor.
Time Frame: 9 years(MAX)
Population: The safety analysis population consists of the cases that satisfy the cases conditions and in whom administration of this drugs was confirmed.
Measure: Number; unit: participants
Groups:
- Azithromycin With Concomitant Drugs: Participants with concomitant drugs who taking Azithromycin for Prophylaxis according to Japanese Package Insert.
- Azithromycin Without Concomitant Drugs: Participants without concomitant drugs who taking Azithromycin for Prophylaxis according to Japanese Package Insert.
Arm/Group | Azithromycin With Concomitant Drugs | Azithromycin Without Concomitant Drugs
Number analyzed (Participants) | 387 | 4
participants | 73 | 0
Statistical Analysis 1: Comparison: Azithromycin With Concomitant Drugs vs Azithromycin Without Concomitant Drugs; The risk factor tested was "concomitant drugs". The null hypothesis is there is no difference between "with and without concomitant drugs " in the frequency of Treatment Related Adverse Events(TRAEs); Test type: Superiority or Other; p = 1.000, Fisher Exact

6. Primary Outcome: Risk Factors for the Frequency of Treatment Related Adverse Events -Renal Dysfunction (Prophylaxis).
Description: Number of participants with Treatment Related Adverse Events(TRAEs) of Azithromycin to determine whether with or without renal dysfunction is significant risk factor.
Time Frame: 9 years(MAX)
Population: as for outcome 3
Measure: Number; unit: participants
Groups:
- Azithromycin With Renal Dysfunction: Participants with renal dysfunction who taking Azithromycin for Prophylaxis according to Japanese Package Insert.
- Azithromycin Without Renal Dysfunction: Participants without renal dysfunction who taking Azithromycin for Prophylaxis according to Japanese Package Insert.
Arm/Group | Azithromycin With Renal Dysfunction | Azithromycin Without Renal Dysfunction
Number analyzed (Participants) | 13 | 378
participants | 2 | 71
Statistical Analysis 1: Comparison: Azithromycin With Renal Dysfunction vs Azithromycin Without Renal Dysfunction; The risk factor tested was "Renal Dysfunction". The null hypothesis is there is no difference between "with and without renal dysfunction " in the frequency of Treatment Related Adverse Events(TRAEs); Test type: Superiority or Other; p = 1.000, Fisher Exact

7. Primary Outcome: Risk Factors for the Frequency of Treatment Related Adverse Events -Allergies (Prophylaxis).
Description: Number of participants with Treatment Related Adverse Events(TRAEs) of Azithromycin to determine whether with or without allergies is significant risk factor.
Time Frame: 9 years(MAX)
Population: as for outcome 3
Measure: Number; unit: participants
Groups:
- Azithromycin With Allergies: Participants with allergies who taking Azithromycin for Prophylaxis according to Japanese Package Insert.
- Azithromycin Without Allergies: Participants without allergies who taking Azithromycin for Prophylaxis according to Japanese Package Insert.
Arm/Group | Azithromycin With Allergies | Azithromycin Without Allergies
Number analyzed (Participants) | 108 | 226
participants | 28 | 33
Statistical Analysis 1: Comparison: Azithromycin With Allergies vs Azithromycin Without Allergies; The risk factor tested was "Allergies". The null hypothesis is there is no difference between "with and without allergies" in the frequency of Treatment Related Adverse Events(TRAEs); Test type: Superiority or Other; p = 0.015, Fisher Exact

8. Primary Outcome: Risk Factors for the Frequency of Treatment Related Adverse Events -Age (Treatment).
Description: as for outcome 3
Time Frame: 9 years(MAX)
Population: as for outcome 3
Measure: Number; unit: participants
Groups:
- <65 Years: Participants with <65 years who taking Azithromycin for Treatment according to Japanese Package Insert.
- >=65 Years: Participants with >=65 years who taking Azithromycin for Treatment according to Japanese Package Insert.
Arm/Group | <65 Years | >=65 Years
Number analyzed (Participants) | 83 | 1
participants | 10 | 0
Statistical Analysis 1: Comparison: <65 Years vs >=65 Years; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 1.000, Fisher Exact

9. Primary Outcome: Risk Factors for the Frequency of Treatment Related Adverse Events -Gender (Treatment).
Description: as for outcome 4
Time Frame: 9 years(MAX)
Population: as for outcome 3
Measure: Number; unit: participants
Groups:
- Male: Male Participants taking Azithromycin for Treatment according to Japanese Package Insert.
- Female: Female Participants taking Azithromycin for Treatment according to Japanese Package Insert.
Arm/Group | Male | Female
Number analyzed (Participants) | 75 | 9
participants | 8 | 2
Statistical Analysis 1: Comparison: Male vs Female; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.290, Fisher Exact

10. Primary Outcome: Risk Factors for the Frequency of Treatment Related Adverse Events -Renal Dysfunction (Treatment).
Description: as for outcome 6
Time Frame: 9 years(MAX)
Population: as for outcome 3
Measure: Number; unit: participants
Groups:
- Azithromycin With Renal Dysfunction: Participants with renal dysfunction who taking Azithromycin for Treatment according to Japanese Package Insert.
- Azithromycin Without Renal Dysfunction: Participants without renal dysfunction who taking Azithromycin for Treatment according to Japanese Package Insert.
Arm/Group | Azithromycin With Renal Dysfunction | Azithromycin Without Renal Dysfunction
Number analyzed (Participants) | 7 | 77
participants | 4 | 6
Statistical Analysis 1: Comparison: Azithromycin With Renal Dysfunction vs Azithromycin Without Renal Dysfunction; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.003, Fisher Exact

11. Primary Outcome: Risk Factors for the Frequency of Treatment Related Adverse Events -Allergies (Treatment).
Description: as for outcome 7
Time Frame: 9 years(MAX)
Population: as for outcome 3
Measure: Number; unit: participants
Groups:
- Azithromycin With Allergies: Participants with allergies who taking Azithromycin for Treatment according to Japanese Package Insert.
- Azithromycin Without Allergies: Participants without allergies who taking Azithromycin for Treatment according to Japanese Package Insert.
Arm/Group | Azithromycin With Allergies | Azithromycin Without Allergies
Number analyzed (Participants) | 19 | 56
participants | 3 | 7
Statistical Analysis 1: Comparison: Azithromycin With Allergies vs Azithromycin Without Allergies; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.707, Fisher Exact

12. Secondary Outcome: Number of Participants That Responded to Azithromycin Treatment.
Description: The physician performed efficacy evaluations at the end of the observation period (or the time of discontinuing administration), compared with the data before the start of administration of this drug, and entered the results.
Time Frame: 9 years(MAX)
Population: The efficacy analysis population basically consists of the evaluable cases in accordance with the separately prepared analysis plan (cases judged to have been evaluated appropriately).
Measure: Number; unit: participants
Arm/Group | Azithromycin for Treatment
Number analyzed (Participants) | 64
participants | 51

13. Secondary Outcome: Number of Participants Prevented by Azithromycin Treatment.
Description: as for outcome 12
Time Frame: 9 years(MAX)
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Azithromycin for Prophylaxis
Number analyzed (Participants) | 390
participants | 375

ADVERSE EVENTS:
Description: The frequency of treatment related advers events during the study.
Arm/Group | Azithromycin for Prophylaxis | Azithromycin for Treatment
Serious Adverse Events (participants affected / at risk) | 11/391 | 4/84
Other Adverse Events (participants affected / at risk) | 62/391 | 6/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin for Prophylaxis (N=391) | Azithromycin for Treatment (N=84)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 (0) | 1 (1)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (3) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin for Prophylaxis (N=391) | Azithromycin for Treatment (N=84)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 1 (1)
Duodenal ulcer (General disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 5 (5) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 5 (5) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Sexual dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 4 (4) | 1 (1)
Platelet count decreased (Investigations) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Beta 2 microglobulin urine increased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.